CLINICAL TRIAL: NCT05322252
Title: Simultaneous Mifepristone and Misoprostol Versus Misoprostol Alone for Induction of Labor of Nonviable Second Trimester Pregnancy: a Pilot Randomized Controlled Trial
Acronym: MIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Katherine Hollister Bligard, Maternal-Fetal Medicine Fellow, Washington University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202202144
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-04

CONDITIONS: Abortion, Second Trimester; PPROM; Rupture, Spontaneous; Fetal Demise; Fetal Death; Fetal Demise From Miscarriage; Fetal Death Before 22 Weeks With Retention of Dead Fetus; Pregnancy Loss; Pregnancy Complications
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Rupture, Spontaneous; Fetal Death; Pregnancy Complications | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simulatenous mifepristone and misoprostol (Experimental): Participants will receive a dose of 200mg oral mifepristone at time of induction with misoprostol
  Interventions: Drug: Mifepristone; Drug: Misoprostol
- Misoprostol alone (Active Comparator): Participants will have labor induced with misoprostol alone
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — 200mg orally
  Arms: Simulatenous mifepristone and misoprostol
Drug: Misoprostol — Per clinician

SUMMARY:
When time allows, administration of mifepristone prior to second trimester induction of labor decreases total labor time. However, in the setting of many pregnancy complications, decreasing time from diagnosis of nonviable pregnancy to delivery is of utmost importance to decrease risk of maternal complications. Previous data has shown that total abortion time is longer in the group receiving mifepristone owing to the delay between mifepristone administration and initiation of misoprostol induction of labor. Thus, the investigators aim to investigate whether simultaneous mifepristone and misoprostol has benefits over misoprostol alone when labor induction of a nonviable second trimester cannot be delayed.

DETAILED DESCRIPTION:
Up to 3% of pregnancies in the second trimester are nonviable and require delivery due to myriad complications including stillbirth, preterm prelabor rupture of membranes (PPROM) at a previable gestational age, fetal anomalies, or risk to maternal life. Stillbirth complicates in 1 in 160 deliveries, with over half of these occurring in the second trimester. Additionally, the rate of preterm previable PPROM is estimated to complicate up to 1% of all pregnancies. The rate of neonatal survival after previable PPROM after expectant management is reported to be as low as 20% due to complications from premature delivery, inadequate fetal lung development, and infectious complications. On the other hand, pregnancy continuation in the setting of previable PPROM increases maternal risk of bleeding, infection, sepsis, and even death. Most fetal anomalies including those that are lethal or associated with severe morbidity are diagnosed after 20 weeks' gestation which is the standard time for the ultrasound assessment of fetal anatomy. Lastly, at any time in pregnancy maternal medical complications can arise or worsen that make continuation of pregnancy contraindicated due to threat to maternal life. Patients in these and other complex situations are counseled on options for the pregnancy, and many make the decision to proceed with induction of labor with the understanding that the fetus will not survive to hospital discharge.

The standard of care for labor induction of a nonviable second trimester pregnancy is the use of misoprostol. However, mifepristone's adjunctive use to shorter time to delivery in the second trimester has become a topic of interest. Mifepristone, also known as RU-486, is a well-tolerated competitive progesterone receptor antagonist. Data has demonstrated the safety and efficacy of mifepristone administration followed by misoprostol 1-2 days later in medical management of first-trimester pregnancy loss and in first-trimester medication abortion. Newer data suggests that mifepristone administration prior to labor induction with misoprostol in nonviable pregnancies decreases total time in labor, with optimal time interval between mifepristone and misoprostol administration thought to be 24-48 hours. However, when considering the time from first medication administration to delivery, the time is longer in those patients receiving mifepristone, owing to the delay from mifepristone administration to induction of labor. A retrospective review of our patients undergoing induction of labor for nonviable second trimester pregnancies from 2018 to 2021 revealed an average length of time from first medication administration to placental delivery of 13.8 hours in patients receiving misoprostol alone, compared to 43.3 hours in those receiving mifepristone at least 24 hours prior to induction of labor (p<0.01). In the setting of many second trimester pregnancies requiring delivery, shortening the time from diagnosis of pregnancy complication and initiation of labor induction to delivery is of utmost importance to decrease the risk of maternal morbidity with a continuing pregnancy. Currently, given need to expedite delivery, these patients are generally induced with misoprostol without adjunctive mifepristone as mifepristone's effectiveness given concurrently with labor induction is unknown. However, pharmacokinetic studies of mifepristone demonstrate that peak concentrations are reached within 60-120 minutes and remain elevated for at least 48 hours, thus it is reasonable to suspect that mifepristone administered at the initiation of labor induction could offer some benefit to patients needing urgent delivery. Thus, the investigators are conducting a randomized controlled trial investigating the utility of simultaneous mifepristone administration at the time of complicated nonviable labor induction with misoprostol in the second trimester.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* 14 and 28 weeks' gestation
* Singleton gestation
* Nonviable fetus (i.e. fetal demise or previable gestational age/weight or lethal fetal anomaly)
* Requires induction of labor
* If fetal cardiac motion, abortion being performed for medical emergency per MO laws and consents completed

Exclusion Criteria:

* Contraindication to mifepristone
* Plan for surgical evacuation of uterus
* Contraindication to vaginal delivery
* Plan to initiate induction with any medication or device except misoprostol
* Declines participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Delivery within 12 hours | 12 hours
  Delivery of fetus and placenta

SECONDARY OUTCOMES:
Delivery within 24 hours | 24 hours
  Delivery of fetus and placenta
Time to delivery | During admission
  Time from misoprostol to delivery of fetus and placenta
Failed induction of labor | During admission
  Need for surgical evacuation of fetus via dilation and evacuation
Retained placenta | During admission
  Need for surgical evacuation of placenta or membranes via dilation and curettage or manual vacuum aspiration
Diagnosis of clinical chorioamnionitis | During admission
  Infection within the uterus during labor induction as diagnosed by obstetrician
Postpartum hemorrhage | During admission
  Blood loss of greater than 1000mL or with hemodynamic instability

OTHER OUTCOMES:
Pregnancy related readmission within 30 days | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided